CLINICAL TRIAL: NCT00636428
Title: Clinical Trial of Oral Midazolam in Pediatric Endoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tabriz University (Other)
Responsible Party: Alireza Javadzadeh, Tabriz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 85-24
Record Dates: First submitted 2008-03-07; First posted 2008-03-14 (Estimated); Last update posted 2008-04-11 (Estimated); Status verified 2008-04

CONDITIONS: Endoscopy
Keywords: endoscopy; Midazolam; pediatric; sedation; comfort
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Oral midazolam
  Interventions: Drug: Midazolam
- 2 (Active Comparator): IV Midazolam
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Midazolam — oral midazolam, was prepared into a final solution (2.5 mg/mL) from injectable midazolam hydrochloride and a orange flavored syrup. For preparation, midazolam injection (5 mg/mL) was diluted 1:1 with the flavored syrup.

SUMMARY:
The objective of our study was to compare the safety and efficacy of oral midazolam during pediatric endoscopy.

DETAILED DESCRIPTION:
Although gastrointestinal endoscopy is widely accepted as fundamental to the diagnosis and treatment of digestive disorders in children, considerable controversy and practice differences persist with respect to the methods and agents used to achieve optimal endoscopic sedation.

Comparison:oral midazolam vs midazolam IV in sedation and comfort scale of pediatric endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* All of patients scheduled for endoscopy participated in the study.

Exclusion Criteria:

Exclusion criteria were as follows:

* Children younger than 3 years;
* Children with significant neurological disability;
* Children with a history of allergies to benzodiazepines, or to their components;
* Children with metabolic, cardiac or renal disease; children with previous - Complications to IV sedation;
* Children with respiratory distress
* Age under 1 mo and bigger than 17y
* History of erythromycin used in 4 week ago

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2007-03; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
efficacy and safety of endoscopy in children with used midazolam

SECONDARY OUTCOMES:
The level of sedation
patient complications, ease of performing the procedure, time of preparation, time for recovery

CONTACTS AND LOCATIONS:
Overall Officials: mandana Rafeey, Dr, Study Chair — liver &Gastrointestinal Research center of tabriz medical university; Mandana Rafeey, Dr, Study Chair — tabriz medical university
Locations (1):
- Liver &Gastrointestinal Research center of tabriz medical university, Tabriz, East Azarbijan, Iran